CLINICAL TRIAL: NCT06199388
Title: Development and Validation of a Deep Learning-Based Survival Prediction Model for Pediatric Glioma Patients: A Retrospective Study Using the SEER Database and Chinese Data
Status: Completed | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDLL-202312-05
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SEER database: The model was trained using the Surveillance, Epidemiology, and End Results (SEER) Registry database. To identify specific tumor types, the International Classification of Diseases for Oncology, 3rd Edition codes (ICD-O-3) were used, including codes 9450, 9394, 9421, 9384, 9383, 9424, 9400, 9420, 9410, 9411, 9380, 9382, 9391, 9393, 9390, 9401, 9381, 9451, 9440, 9441, 9442, 9430, and 9380, covering astrocytic tumors, oligodendroglia tumors, oligoastrocytic tumors, ependymal tumors, and other gliomas. Inclusion criteria comprised all primary brain tumors (C71.0-C71.9, C72.3, C72.8, C75.3) diagnosed between 2000 and 2018, among patients under 21 years old, and meeting the third edition of the ICD-O-3 classification. Only patients with available survival time were included, and those with unknown or missing clinical features were excluded.
  Interventions: Other: Survival state
- Chinese cohort: To assess the generalizability of the final model, an external validation cohort from China was used. This cohort consisted of 258 pediatric glioma patients diagnosed at Tangdu Hospital in Xi'an, China, between January 2010 and December 2018. These patients had complete clinical data and comprehensive follow-up records.
  Interventions: Other: Survival state

INTERVENTIONS:
Other: Survival state — We recorded clinically relevant information and survival status of pediatric glioma patients

SUMMARY:
Accurately predicting the survival of pediatric glioma patients is crucial for informed clinical decision-making and selecting appropriate treatment strategies. However, there is a lack of prognostic models specifically tailored for pediatric glioma patients. This study aimed to address this gap by developing a time-dependent deep learning model to aid physicians in making more accurate prognostic assessments and treatment decisions.

DETAILED DESCRIPTION:
This retrospective study focuses on survival prediction in pediatric glioma patients using a population-based approach. The model was trained using the Surveillance, Epidemiology, and End Results (SEER) Registry database. To identify specific tumor types, the International Classification of Diseases for Oncology, 3rd Edition codes (ICD-O-3) were used, including codes 9450, 9394, 9421, 9384, 9383, 9424, 9400, 9420, 9410, 9411, 9380, 9382, 9391, 9393, 9390, 9401, 9381, 9451, 9440, 9441, 9442, 9430, and 9380, covering astrocytic tumors, oligodendroglia tumors, oligoastrocytic tumors, ependymal tumors, and other gliomas. Inclusion criteria comprised all primary brain tumors (C71.0-C71.9, C72.3, C72.8, C75.3) diagnosed between 2000 and 2018, among patients under 21 years old, and meeting the third edition of the ICD-O-3 classification. Only patients with available survival time were included, and those with unknown or missing clinical features were excluded. This cohort consisted of 258 pediatric glioma patients diagnosed at Tangdu Hospital in Xi'an, China, between January 2010 and December 2018. These patients had complete clinical data and comprehensive follow-up records.

ELIGIBILITY:
Inclusion Criteria:

* To identify specific tumor types, the International Classification of Diseases for Oncology, 3rd Edition codes (ICD-O-3) were used, including codes 9450, 9394, 9421, 9384, 9383, 9424, 9400, 9420, 9410, 9411, 9380, 9382, 9391, 9393, 9390, 9401, 9381, 9451, 9440, 9441, 9442, 9430, and 9380, covering astrocytic tumors, oligodendroglia tumors, oligoastrocytic tumors, ependymal tumors, and other gliomas. Inclusion criteria comprised all primary brain tumors (C71.0-C71.9, C72.3, C72.8, C75.3) diagnosed, among patients under 21 years old, and meeting the third edition of the ICD-O-3 classification.

Exclusion Criteria:

* Only patients with available survival time were included, and those with unknown or missing clinical features were excluded.

Max Age: 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: the US Surveillance, Epidemiology, and End Results (SEER) between January 2000 and December 2018 and a Chinese registry (The Tangdu Hospital of the Fourth Military Medical Universitye) between January 2010 and December 2018
Sampling Method: Probability Sample
Enrollment: 9532 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
overall survival | 2000.01-2018.12
  The primary outcome was overall survival (OS), which was defined as the time interval from the pediatric glioma diagnosis until death or the end of follow-up in SEER registry
overall survival | 2010.01-2018.12
  The primary outcome was overall survival (OS), which was defined as the time interval from the pediatric glioma diagnosis until death or the end of follow-up in Chinese registry

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No
The data involves the relevant personal privacy information of the patient

REFERENCES:
- [Result] Thomas L, Li F, Pencina M. Using Propensity Score Methods to Create Target Populations in Observational Clinical Research. JAMA. 2020 Feb 4;323(5):466-467. doi: 10.1001/jama.2019.21558. No abstract available. PMID 31922529
- [Result] Doll KM, Rademaker A, Sosa JA. Practical Guide to Surgical Data Sets: Surveillance, Epidemiology, and End Results (SEER) Database. JAMA Surg. 2018 Jun 1;153(6):588-589. doi: 10.1001/jamasurg.2018.0501. No abstract available. PMID 29617544